CLINICAL TRIAL: NCT05371015
Title: Quadratus Lumborum Block Reduced Postpartum Uterine Pain After Virginal Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202102060A3
Record Dates: First submitted 2022-04-05; First posted 2022-05-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2022-02

CONDITIONS: Quadratus Lumborum Nerve Block; Postpartum Cramping; Vaginal Delivery
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Fifty subjects were randomly assigned to the quadratus lumborum nerve block group with injection of local anesthetic (Ropivacaine), and another 50 subjects were assigned to the quadratus lumborum nerve block with normal saline injection. The total number of subjects involved is one hundred.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After the computer program (SAS® 9.4) generates the groups of subjects in random order, a third-party person who is not the research team will put the groups into envelopes numbered one to one hundred in sequence. Which group the subjects will be assigned to will not be known to members of the research team until the trial is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadratus lumborum nerve block group with injection of local anesthetic (Ropivacaine) (Experimental): The subjects would have quadratus lumborum nerve block group with injection of local anesthetic (Ropivacaine) after vaginal delivery.
  Interventions: Procedure: quadratus lumborum nerve block (ropivacaine )
- quadratus lumborum nerve block with normal saline (Placebo Comparator): The subjects would have quadratus lumborum nerve block with normal saline after vaginal delivery.
  Interventions: Procedure: quadratus lumborum nerve block (normal saline)

INTERVENTIONS:
Procedure: quadratus lumborum nerve block (ropivacaine ) — Echo guided quadratus lumborum nerve block with ropivacaine
  Other Names: QLB
  Arms: quadratus lumborum nerve block group with injection of local anesthetic (Ropivacaine)
Procedure: quadratus lumborum nerve block (normal saline) — Echo guided quadratus lumborum nerve block with normal saline
  Other Names: QLB
  Arms: quadratus lumborum nerve block with normal saline

SUMMARY:
With the continuous advancement of ultrasonic technology, nerve block in which drugs are injected into the periphery of the target nerve through ultrasonic guidance has become the mainstream method for postoperative pain control. The quadratus lumborum nerve block has been effectively and safely used in abdominal surgery (such as laparotomy, caesarean section, etc.), effectively reducing postoperative wounds and visceral pain. There is no research on the use of quadratus lumborum nerve block to control the pain of natural postpartum uterine contractions in the current literature, so the purpose of this experiment is to explore whether the quadratus lumborum nerve block can effectively reduce the pain of uterine contractions after vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Females over twenty years of age
* Maternal vaginal delivery
* Postpartum moderate to severe pain with uterine contractions (Numerical Pain Scale (NRS) ≥ 4 points) after delivery.
* Subject's consent signed by the subject

Exclusion Criteria:

* Severe coagulation abnormalities (PLT<100000、INR>1.2、PT>13)
* Infection of the epidermis at the anticipated relevant site of injection
* Allergy to local anesthetics
* Allergy to or abuse of pain control medications
* Episiotomy is more painful than uterine contractions
* Inability to cooperate with associated pain assessment
* Body Mass Index (BMI) ≧ 35 kg/m2

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female had maternal vaginal delivery
Enrollment: 66 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Pain associated with uterine contractions | Right before intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 1 hour after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 6 hours after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 12 hours after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 24 hours after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 36 hours after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]
Pain associated with uterine contractions | 48 hours after intervention
  Grading with Numerical Pain Scale [0 (no pain at all) to 10 (worst imaginable pain)] and Visual Analogue Scale [mark a position between 0 (no pain at all) to 10 (worst imaginable pain)]

OTHER OUTCOMES:
Edinburgh Postnatal Depression Scale | Right before intervention
  Edinburgh Postnatal Depression Scale 10-item (ranging from 0 to 30, possible depression > 10)
Pittsburgh sleep quality index | Right before intervention
  Pittsburgh sleep quality index (ranging from 0 to 21, where lower scores denote a healthier sleep quality)
Modified Fatigue Symptoms Checklist | Right before intervention
  Modified Fatigue Symptoms Checklist (ranging from 0 to 40, where higher scores mean more exhausted physical and mental status)
Postpartum Perceived Stress Scale | Right before intervention
  Postpartum Perceived Stress Scale - 14 items (range from 0 to 70 with higher scores indicating higher perceived stress)
Edinburgh Postnatal Depression Scale | 48 hours after intervention
  Edinburgh Postnatal Depression Scale 10-item (from 0 to 30, possible depression > 10)
Pittsburgh sleep quality index | 48 hours after intervention
  Pittsburgh sleep quality index Modified Fatigue Symptoms Checklis (ranging from 0 to 21, where lower scores denote a healthier sleep quality)
Modified Fatigue Symptoms Checklist | 48 hours after intervention
  Modified Fatigue Symptoms Checklist (ranging from 0 to 40, where higher scores mean more exhausted physical and mental status)
Postpartum Perceived Stress Scale | 48 hours after intervention
  Postpartum Perceived Stress Scale - 14 items (range from 0 to 70 with higher scores indicating higher perceived stress)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital (Linkou), Taoyuan, Taiwan